CLINICAL TRIAL: NCT04209374
Title: Etude de Cohorte Observationnelle Rétrospective SYMBOL CUP 1
Brief Title: Retrospective Observational Cohort Study of SYMBOL CUP DM 1
Acronym: SYMCOR-1
Status: Completed | Type: Observational
Sponsor: Dedienne Sante S.A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: SYMCOR-1
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: primary total hip arthroplasty; hemispherical dual-mobility acetabular cup; safety; efficacy; implant survival; prosthetic dislocation; Harris hip score HHS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HMB-DMR-HA: Primary total hip arthroplasty with hemispherical dual-mobility acetabular cup
  Interventions: Device: THA with SYMBOL CUP DM HA

INTERVENTIONS:
Device: THA with SYMBOL CUP DM HA

SUMMARY:
This is a single-center retrospective observational cohort study of consecutively operated patients who underwent primary total hip arthroplasty with a SYMBOL CUP DM HA hemispherical dual mobility acetabular implant. The purpose of this study is to estimate the safety and efficacy of that implant at two-year follow-up.

DETAILED DESCRIPTION:
Description according to PICOS framework:

Patients:

- Adult men and women requiring a primary total hip arthroplasty

Intervention:

- Primary THA with SYMBOL CUP DM HA hemispherical dual mobility acetabular implant.

Comparator: None

Outcomes:

* Safety 1: Implant survival over 2-year follow-up.
* Safety 2: All adverse events, with focus on implant dislocation, infections, revision surgery
* Efficacy 1: Harris Hip Score (HHS) at baseline and 1-year follow-up.
* Efficacy 2: Modified HHS consisting of pain + functional subscores at baseline, 1-year and 2-year follow-ups.
* Efficacy 2: Devane score at baseline, 1-year and 2-year follow-ups.
* Efficacy 3: Charnley classification at baseline, 1-year and 2-year follow-ups.

Study design:

* single-center retrospective observational cohort study of consecutively operated patients who underwent primary total hip arthroplasty 2 years prior to study start.
* Prospective 2-year follow-up letter and phone questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients with total hip implant using hemispheric dual-mobility SYMBOL CUP DM HA
* Operation performed by the primary investigator
* Delay between index operation and March 1 2018 has reached 2 years

Exclusion Criteria:

* patient refusal to participate in the study
* minors (age < 18 years)
* patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exhaustive recruitment of patients meeting inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Implant survival: Ratio of the number of participants alive with the complete index hip prosthesis in position at 2-year follow-up, over their initial numberprosthesis in position at 2-year follow-up, over their initial number. | 2 years as of index operation
  This is the ratio of the number of participants who are alive with the complete index hip prosthesis in position at a given follow-up time (numerator) over the initial number of those participants from the date they received the index hip prosthesis (denominator). The cumulative ratio is recalculated at each event using the Kaplan-Meier method from the date of each participant index operation through the date of each participant's death or prosthetic removal surgery or loss-to-follow-up or last assessment alive with the hip prosthesis in place. The longest duration between the index operation and the final assessment is 2 years.

SECONDARY OUTCOMES:
Number of patients with one or several post-operative adverse events and count of each Serious adverse event and aggregate count of adverse events | 2 years as of index operation
  All serious post-operative adverse events are taken into account including implant dislocation, infections, revision surgery
Harris Hip Score (HHS) at baseline and 1-year follow-up | 1 year as of index operation
  The score is measured at each assessment in each patient. The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments
The modified Harris Hip Score (modified HHS) at baseline, 1-year and 2-year follow-up | 2 years as of index operation
  The modified Harris Hip Score (modified HHS) is the sum of pain subscore and functional subscore of the Harris Hip Score. The score is measured at each assessment in each patient. The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments
Devane classification at baseline, 1-year and 2-year follow-up. | 2 years as of index operation
  The class is measured at each assessment in each patient. The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments
Charnley classification at baseline, 1-year and 2-year follow-up. | 2 years as of index operation
  The class is measured at each assessment in each patient. The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bonin, M.D., Principal Investigator — Lyon Ortho Clinic - Clinique de la Sauvegarde
Locations (1):
- Lyon Ortho Clinic - Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No